CLINICAL TRIAL: NCT03613844
Title: The Delivery of Essential Fatty Acids to the Brain
Brief Title: DHA Brain Delivery Trial
Acronym: PreventE4
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: Huntington Medical Research Institutes (Other); National Institute on Aging (NIA) (NIH); Alzheimer's Drug Discovery Foundation (Other)
Responsible Party: Principal Investigator, Hussein Yassine, Assistant Professor, University of Southern California
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: HS-18-00291/00984; R01AG054434 (NIH); GC-201711-2014197 (Other Grant/Funding Number: Alzheimer's Drug Discovery Foundation)
Record Dates: First submitted 2018-07-11; First posted 2018-08-03 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Brain DHA Delivery and Alzheimer's Disease Risk
Keywords: Alzheimer's disease; Docosahexaenoic Acids; Apolipoprotein E4
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: double blind and randomized placebo controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DHA (Experimental): oral DHA supplementation at 2 grams per day
  Interventions: Drug: DHA
- Placebo (Placebo Comparator): Placebo for DHA
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DHA — DHA supplementation
  Arms: DHA
Drug: Placebo — Placebo for DHA
  Arms: Placebo

SUMMARY:
Carrying the APOE ɛ4 allele is the strongest genetic risk factor for developing Alzheimer's disease. The goal of this project is to identify whether carrying the APOE ɛ4 allele is associated with reduced delivery of DHA to the brain. This information will help us identify the target population that could benefit from DHA supplementation to prevent cognitive decline.

DETAILED DESCRIPTION:
The Brain DHA Delivery Trial will examine the effect of APOE genotype on the changes of cerebrospinal fluid (CSF) DHA to Arachidonic acid (AA) ratio in 184 cognitively healthy older individuals in response to DHA supplementation. Randomized clinical trials have yielded mixed results on the effect DHA supplementation on cognitive outcomes. This study asks the critical question of whether DHA gets into the brain in sufficient amounts after supplementation, and whether APOE genotype affects brain penetrance.

This trial will also test the effect of DHA supplementation on changes in brain structural and functional connectivity assessed by MRI, and changes in cognition after two years of supplementation in all 368 participants.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥ 55 and ≤ 80
* At least one dementia risk factor (obesity, education years, hypertension, hyperlipidemia)
* Mini-Mental State Examination (MMSE) ≥ 25
* Logical Memory II delayed recall score ≥ 6 and ≤ 18 .

Exclusion Criteria:

* Diagnosis of dementia as assessed by the investigator
* Use of omega-3 preparations in the last 3 months
* > 200 mg/day of DHA consumption using a validated questionnaire
* Use of donepezil, rivastigmine, galantamine and/or memantine
* Alcohol or drug abuse
* A concomitant serious disease such as active cancer treatment or HIV.
* Participation in a clinical trial in the last 30 days
* Use of anticoagulants such as Plavix or Coumadin or the newer generation blood thinners.

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 365 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

PRIMARY OUTCOMES:
change in cerebrospinal fluid fatty acid levels after the intervention in 184 subjects | 6 months
  cerebrospinal fluid fatty acids assessed by mass spectrometry

OTHER OUTCOMES:
Change in functional connectivity using resting state functional MRI in all 368 participants | 2 years
  Functional Connectivity
Change in structural connectivity using MRI in all 368 participants | 2 years
  Structural connectivity
Change in cognitive measures using the Neuropsychological Outcomes (RBANS) in all 368 participants | 2 years
  RBANS battery

CONTACTS AND LOCATIONS:
Overall Officials: Hussein Yassine, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Keck School of Medicine, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
available by request to study principal investigator and after approval by study committee.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: within 1 year after study publication

REFERENCES:
- [Background] Yassine HN, Braskie MN, Mack WJ, Castor KJ, Fonteh AN, Schneider LS, Harrington MG, Chui HC. Association of Docosahexaenoic Acid Supplementation With Alzheimer Disease Stage in Apolipoprotein E epsilon4 Carriers: A Review. JAMA Neurol. 2017 Mar 1;74(3):339-347. doi: 10.1001/jamaneurol.2016.4899. PMID 28114437
- [Derived] Yassine HN, Arellanes IC, Mazmanian A, De La Cruz L, Martinez J, Contreras L, Kono N, Liu BS, Badie D, Bantugan MA, Grindon A, Urich T, D'Orazio L, Emmanuel BA, Chui HC, Mack WJ, Harrington MG, Braskie MN, Schneider LS. Baseline Findings of PreventE4: A Double-Blind Placebo Controlled Clinical Trial Testing High Dose DHA in APOE4 Carriers before the Onset of Dementia. J Prev Alzheimers Dis. 2023;10(4):810-820. doi: 10.14283/jpad.2023.77. PMID 37874103